CLINICAL TRIAL: NCT00559260
Title: Evaluation of Cardiorespiratory Events in Subjects Undergoing an Upper and/or Lower Endoscopy Under Current Sedation Practices While Being Passively Monitored
Brief Title: Evaluation of Cardiorespiratory Events in Subjects Undergoing an Upper and/or Lower Endoscopy Under Current Sedation Practices
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Other Study IDs: CI-02-0004
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Sedation for Non-Emergent Upper and/or Lower Endoscopy
MeSH Terms: interventions — Oximetry; Electrocardiography

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Passive monitoring with pulse-oximetry, NIBP and ECG

SUMMARY:
This is a 300 subject prospective study to assess cardiorespiratory events associated with current practice sedation (150 subjects; opioid + benzodiazepine) versus anesthesia provider sedation (150 subjects; propofol) for upper and/or lower endoscopy.

ELIGIBILITY:
Inclusion Criteria:adult

* (>=18 years),ASA I-III, non-emergent upper and/or lower endoscopy

Exclusion Criteria:

* Emergent indications for upper and/or lower endoscopy (i.e., acute hemorrhage, cholangitis)
* Baseline respiratory rate of < 6 breaths per minute
* Baseline hypotension (systolic blood pressure < 90 mm Hg)
* Baseline arterial oxygen saturation < 90% on room air
* Baseline bradycardia: heart rate < 50 beats per minute
* Baseline tachycardia: heart rate > 110 beats per minute
* Allergy or inability to tolerate any of the sedatives or analgesics to be administered during the procedure
* Inability to squeeze the Automated Responsiveness Test hand piece (last 50 subjects only)
* Significant hearing impairment
* Actively abusing alcohol, opioids, benzodiazapines or sedatives, or other drugs
* Are considered tolerant to opioids, benzodiazapines and/or other sedatives through prescription.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Philip Miner, MD, Principal Investigator — Oklahoma Foundation for Digestive Research
Locations (1):
- Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma, United States